CLINICAL TRIAL: NCT02363387
Title: Suppression of HIV 1 RNA in People Living With HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00044740; R01AI117065 (NIH)
Record Dates: First submitted 2015-02-05; First posted 2015-02-16 (Estimated); Results first posted 2023-04-24 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: HIV
Keywords: HIV; antiretroviral medications; incentives

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Incentive Group (Experimental): Incentive group participants will receive the standard HIV medical care offered in their clinic. In addition, Incentive group participants will receive incentives for viral suppression. These incentives will be presented if the participants maintain suppressed and undetectable viral loads. The incentive program will employ high magnitude incentives, provide incentives for decreases in viral load early in treatment before a patient's viral load has reached undetectable levels, arrange frequent incentives early in treatment and reduce the frequency of incentives as participants achieve progressively longer periods of viral load suppression, arrange a schedule of escalating incentives for sustained suppression of viral load, and the intervention will be maintained for two years.
  Interventions: Behavioral: Incentives for Viral Suppression; Behavioral: Standard HIV Medical Care
- Usual Care Group (Other): Usual Care Control participants will receive the standard HIV medical care offered in their clinic.
  Interventions: Behavioral: Standard HIV Medical Care

INTERVENTIONS:
Behavioral: Incentives for Viral Suppression — Incentive group participants will receive incentives for maintaining suppressed and undetectable viral loads. The incentive program will employ high magnitude incentives, provide incentives for decreases in viral load early in treatment before a patient's viral load has reached undetectable levels, arrange frequent incentives early in treatment and reduce the frequency of incentives as participants achieve progressively longer periods of viral load suppression, arrange a schedule of escalating incentives for sustained suppression of viral load, and the intervention will be maintained for two years.
  Arms: Incentive Group
Behavioral: Standard HIV Medical Care — The best HIV medical care available in each participant's medical clinic.

SUMMARY:
The investigators propose to evaluate a novel incentive intervention to promote suppression of viral load in people living with HIV that will employ empirically-based parameters that have been proven critical to the effectiveness of incentive interventions. Participants (N = 200) from medical clinics that serve adults living with HIV in Baltimore will be randomly assigned to an Incentive or a Usual Care Control group. Incentive group participants will receive incentives for maintaining suppressed and undetectable viral loads. The incentive program will employ high magnitude incentives, provide incentives for decreases in viral load early in treatment before a patient's viral load has reached undetectable levels, arrange frequent incentives early in treatment and reduce the frequency of incentives as participants achieve progressively longer periods of viral load suppression, arrange a schedule of escalating incentives for sustained suppression of viral load, and the intervention will be maintained for two years. Usual Care Control participants will only receive the standard HIV medical care offered in their clinic. Assessments will be conducted every 3 months throughout the two years of treatment and every 6 months throughout the year following treatment. The primary outcome measure will be the percentage of participants that have undetectable viral loads at the 3-month assessments conducted throughout the 2-year intervention period. Secondary measures will include adherence to HIV care and post-treatment outcomes. The investigators will also assess moderators and mediators of the effects of the incentives on the suppression of viral load, and conduct cost-effectiveness and cost-benefit analyses. If the incentive intervention maintains suppressed viral load and is economically sound, it could be used to improve the health of adults living with HIV, reduce health care costs, and reduce HIV transmission in the community.

DETAILED DESCRIPTION:
Experimental Design. Participants (N = 200) will be randomly assigned to a Usual Care Control group or the Incentive group. A computerized urn randomization procedure (Wei & Lachin, 1988) will be used to balance groups on five baseline characteristics that may influence outcome: (1) Diagnostic and Statistical Manual (DSM) V dependence on cocaine or opiates assessed on the Composite International Diagnostic Interview (CIDI) (Y/N); (2) DSM V alcohol dependence assessed on the CIDI (Y/N); (3) health literacy as assessed on the Test of Functional Health Literacy in Adults (TOFHLA) (score ≤ the rolling median, Y/N); (4) impulsivity as assessed by delay discounting (k value from the raw discounting data for each participant, which is an index of impulsivity (≤ the rolling median of k, Y/N); and (5) depression as assessed by the Beck Depression Inventory (score ≤ the rolling median, Y/N). Participants will be stratified by DSM V cocaine, opiate and alcohol dependence, health literacy, and depression at intake because drug use, health literacy, and depression has each been associated with poor Anti-Retroviral Therapy (ART) adherence. Participants will be stratified based on measures of impulsivity because high levels of impulsivity have been associated with poor health decision making and adverse health behaviors.

Standard HIV Medical Care.

Upon enrollment, participants will be taught about the benefits of ART adherence and the need to maintain nearly perfect adherence. All participants will receive their HIV medical care in their clinic.

Incentive Group.

The Incentive group will receive the novel empirically-based incentive intervention to promote long term suppression of HIV-1 RNA (viral load) being evaluated in this study. The incentive intervention will employ features and parameters that have been shown critically important to promote therapeutic behavior change in drug users and other populations. participants will be taught the details of the incentive program with written instructions and quizzes.

Usual Care Control Group.

Usual Care Control Only participants will receive the standard HIV medical care described above offered in their medical clinic. Participants in this group will not receive added viral load testing, feedback or incentives, beyond the viral load testing conducted as a routine part of their medical care.

ELIGIBILITY:
Inclusion Criteria:

* living with HIV

Exclusion Criteria:

* report current suicidal or homicidal ideation;
* have a severe psychiatric disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2021-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Silverman, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Center for Learning and Health, Johns Hopkins Bayview Medical Campus, 5200 Eastern Ave., Suite W142, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
We will publish the results in a peer-reviewed journal.

REFERENCES:
- [Derived] Novak MD, Holtyn AF, Toegel F, Rodewald AM, Leoutsakos JM, Fingerhood M, Silverman K. Long-Term Effects of Incentives for HIV Viral Suppression: A Randomized Clinical Trial. AIDS Behav. 2024 Feb;28(2):625-635. doi: 10.1007/s10461-023-04249-z. Epub 2023 Dec 20. PMID 38117449

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited participants between 11/1/2015 and 8/30/2017. Participants were recruited in Baltimore from settings that serve people living with HIV and through compensated referrals by participants. Interested individuals completed a brief phone interview. Potentially eligible participants were invited for a full interview.
Groups:
- Incentive Group: Incentive group participants will receive incentives for viral suppression. These incentives will be presented if the participants maintain suppressed and undetectable viral loads. The incentive program will employ high magnitude incentives, provide incentives for decreases in viral load early in treatment before a patient's viral load has reached undetectable levels, arrange frequent incentives early in treatment and reduce the frequency of incentives as participants achieve progressively longer periods of viral load suppression, arrange a schedule of escalating incentives for sustained suppression of viral load, and the intervention will be maintained for two years.
  Incentives for Viral Suppression: Incentive group participants will receive incentives for maintaining suppressed and undetectable viral loads. The incentive program will employ high magnitude incentives, provide incentives for decreases in viral load early in treatment before a patient's viral load has reached undetectable levels, arrange frequent incentives early in treatment and reduce the frequency of incentives as participants achieve progressively longer periods of viral load suppression, arrange a schedule of escalating incentives for sustained suppression of viral load, and the intervention will be maintained for two years.
  Standard HIV Medical Care: The best HIV medical care available in each participant's medical clinic.
Period: Overall Study
Arm/Group | Incentive Group | Usual Care Group
Started | 52 | 50
Completed | 52 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Incentive Group: Incentive group participants will receive the standard HIV medical care offered in their clinic. In addition, Incentive group participants will receive incentives for viral suppression. These incentives will be presented if the participants maintain suppressed and undetectable viral loads.
  Incentives for Viral Suppression: Incentive group participants will receive incentives for maintaining suppressed and undetectable viral loads. The incentive program will employ high magnitude incentives, provide incentives for decreases in viral load early in treatment before a patient's viral load has reached undetectable levels, arrange frequent incentives early in treatment and reduce the frequency of incentives as participants achieve progressively longer periods of viral load suppression, arrange a schedule of escalating incentives for sustained suppression of viral load, and the intervention will be maintained for two years.
  Standard HIV Medical Care: The best HIV medical care available in each participant's medical clinic.
- Total: Total of all reporting groups
Arm/Group | Incentive Group | Usual Care Group | Total
Number analyzed (Participants) | 52 | 50 | 102
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 51 | 50 | 101
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (10) | 47 (9) | 47 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 23 | 47
  Male | 28 | 27 | 55
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 51 | 49 | 100
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 46 | 46 | 92
  White | 4 | 4 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 52 | 50 | 102

OUTCOME MEASURES:

1. Primary Outcome: Undetectable Viral Loads During Treatment
Description: We will assess the percentage of blood samples that have undetectable viral loads (i.e., <200 copies/mL) at the eight 3-month assessments conducted throughout the 2-year intervention evaluation period (Y/N at each assessment).
Time Frame: 2 years
Population: Intent to treat
Measure: Number; unit: percentage of blood samples undetectable
Units Other Than Participants: blood samples
Arm/Group | Incentive Group | Usual Care Group
Number analyzed (Participants) | 52 | 50
Number analyzed (blood samples) | 461 | 400
percentage of blood samples undetectable | 70.4 | 42.5
Statistical Analysis 1: Comparison: Incentive Group vs Usual Care Group; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 7.1, 95% CI 2-sided [2.7 to 18.8]

2. Secondary Outcome: Biologically-verified Adherence to Antiretroviral Medications
Description: We will assess whether the participant maintained consistent ART adherence by conducting qualitative high-resolution mass spectrometry (HRMS) blood tests of 15 antiretroviral medications. Participants will be considered adherent if they test positive for all of their prescribed medications (Y/N at each 3-month assessment).
Time Frame: 2 years
Reporting Status: Not Posted

3. Secondary Outcome: Self-reported Adherence to Antiretroviral Medications
Description: We will assess whether the participant reports maintaining consistent ART adherence by reporting taking >90% of all scheduled doses in the past 30 days (Y/N at each 3-month assessment based on responses on a visual analog scale to assess adherence to antiretroviral medications, see below).
Time Frame: 2 years
Reporting Status: Not Posted

4. Secondary Outcome: Maintaining Prescriptions for Antiretroviral Medications
Description: We will assess the percentage of months that the participant refilled a prescription for antiretroviral medications throughout the 2-year intervention evaluation period (Y/N for each month prior to each 3-month assessment based on timeline follow-back self-report and confirmed by pharmacy records).
Time Frame: 2 years
Reporting Status: Not Posted

5. Secondary Outcome: Retention in HIV Medical Care
Description: We will assess whether the participant attended at least 2 medical visits per year (Y/N each year based on self-report and medical records).
Time Frame: 2 years
Reporting Status: Not Posted

6. Secondary Outcome: Post-intervention Effects
Description: We will assess all primary and secondary outcome measures during the third year of the study after the incentive intervention ends
Time Frame: Year 3
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Incentive Group | Usual Care Group
All-Cause Mortality (participants affected / at risk) | 4/52 | 3/50
Serious Adverse Events (participants affected / at risk) | 10/52 | 1/50
Other Adverse Events (participants affected / at risk) | 0/52 | 0/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Incentive Group (N=52) | Usual Care Group (N=50)
Congestive heart failure (Cardiac disorders) | 0 (0) | 1 (1)
Depression (Nervous system disorders) | 1 (1) | 0 (0)
Hallucinations (Nervous system disorders) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
influenza (Gastrointestinal disorders) | 1 (1) | 0 (0)
Joint pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Kidney failure (General disorders) | 1 (1) | 0 (0)
Pneumonia (General disorders) | 2 (2) | 0 (0)
Psychiatric treatment (Nervous system disorders) | 2 (2) | 0 (0)
Urinary problems (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-14): https://cdn.clinicaltrials.gov/large-docs/87/NCT02363387/Prot_SAP_000.pdf